CLINICAL TRIAL: NCT04456127
Title: Ablative Fractional CO2 Laser Revision for Burn Related Donor Site Scars: A Pilot Randomized Controlled Trial
Brief Title: CO2 Laser Revision for Burn Related Donor Site Scars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-063
Record Dates: First submitted 2020-06-23; First posted 2020-07-02 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Burn Scar; Scar; Skin Graft Scar
Keywords: laser
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: Intra-subject comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care (No Intervention): Scar section does not receive CO2 laser therapy.
- Factional CO2 (Experimental): Scar section receives fractional CO2 laser therapy.
  Interventions: Procedure: Fractional CO2 Laser

INTERVENTIONS:
Procedure: Fractional CO2 Laser — The UltraPulse® fractional ablative CO2 Laser will be employed with the DeepFX™ hand piece. Number of passes and laser settings, including fluency, density, spot size, will be chosen during the time of treatment as determined by the operating surgeon.
  Arms: Factional CO2

SUMMARY:
Scarring from burn wounds remains a chronic and often severe sequela of burn injury. Burn wounds may be left to heal by secondary intention or treated with surgical skin grafting; in both circumstances, significant scars likely result. When surgical skin grafting is employed, skin graft harvest sites ("donor sites") likewise result in clinically significant scars.

This study will have interventional and observational components. Patients will receive the standard fractional ablative CO2 treatments to their scars resulting from burn wounds allowed to heal by secondary intention and/or those treated with skin grafts. These will be prospectively observed for the duration of the study as well as adjacent normal skin. In addition, a donor site that meets inclusion criteria that would not have otherwise received LSR will be identified as a treatment site. Patients with have one half of their donor sites randomized to standard of care (SOC) treatment, which consists of wound dressings, compression therapy, physical and occupational therapies and the other half randomized to SOC + ablative fractional CO2 laser therapy (LSR).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* At least 1 second or third degree burn wound that required treatment with split-thickness skin grafts
* Donor site with at least a 4 x 4 inch surface area
* Able to return to clinical site for treatments and assessments of burn injuries

Exclusion Criteria:

* Pregnancy or nursing
* Oral retinoid medication use within the past 6 months
* Medical history of Ehlers-Danlos syndrome, AIDS
* Nutritional deficiencies in the opinion of the investigator that would affect wound healing
* Wounds complicated by clinically significant infection within past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of Patient and Observer Scar Assessment Scale, VSS, and Delfin Instruments | 2 months
  The primary endpoint will be assessment of control and treatment halves at follow-up evaluation completed 2 months ± 2 weeks after the final laser treatment.
  The change in scale measure from baseline to date of assessment will be used to compare treatment vs control scar halves. This will be calculated and compared using paired t-test with a p-value of 0.05 as the cutoff for significance.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No